CLINICAL TRIAL: NCT00748436
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Examine the Effect of Betahistine on Body Weight in Obese Female Subjects
Brief Title: Efficacy Study of Betahistine on Body Weight in Obese Female Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OBEcure Ltd. (Industry)
Collaborators: International Antiviral Therapy Evaluation Center (Other)
Responsible Party: Yaffa Beck, CEO, OBEcure Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BET207; 2008-001840-38; S51130; ML5059
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Obesity
Keywords: Obese females; Weight loss; Betahistine
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Betahistine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Placebo Comparator): Matching placebo twice a day
  Interventions: Drug: placebo
- B (Experimental): Betahistine 24 mg twice a day (48 mg/day total)
  Interventions: Drug: betahistine dihydrochloride
- C (Experimental): Betahistine 48 mg twice a day (96 mg/day total)
  Interventions: Drug: betahistine dihydrochloride

INTERVENTIONS:
Drug: betahistine dihydrochloride — (24mg tablet Betahistine + placebo tablet) BID per os 12 weeks
  Other Names: Betahistine
  Arms: B
Drug: betahistine dihydrochloride — (24mg tablet Betahistine + 24mg tablet Betahistine) BID per os 12 weeks
  Other Names: Betahistine
  Arms: C
Drug: placebo — (placebo tablet + placebo tablet) BID per os 12 weeks
  Arms: A

SUMMARY:
The purpose of this study is to examine the effect of betahistine on body weight in obese female subjects

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dose finding, multicenter study. The study will consist of 3 treatment groups (48 mg/day, 96 mg/day, and matching placebo). Approximately 180 subjects (60 per treatment group) will be randomized into this 12-week study.

A screening visit will be used to determine subject suitability for inclusion in the trial.

One week after the screening visit subjects who meet all inclusion criteria and none of the exclusion criteria will be randomly assigned to 1 of the following treatment groups:

* Betahistine 24 mg twice a day (BID) (48 mg/day total),
* Betahistine 48 mg BID (96 mg/day total),
* Matching placebo.

All subjects will be prescribed a nutritionally balanced mildly hypocaloric diet. The prescribed diet will contain approximately 30% of calories from fat, 50% of calories from carbohydrates, and 20% of calories from protein. The individual subject's estimated total daily energy expenditure minus 600 kcal will be used to determine each subject's daily caloric intake value during the study. The total daily energy expenditure will be estimated for each subject from the basal energy expenditure multiplied by a correction factor of 1.3 to account for the amount of energy needed in mild to moderate daily activity for obese subjects.

Double-blind treatment will continue for 12 weeks. Study medication (betahistine and/or matching placebo) will be orally administered BID about 1-2 hrs prior to meals (at 10:00 and at 17:00). During this period, 4 additional study visits (at 2, 4, 8, and 12 weeks) will take place.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Female subjects 18 to 50 years of age
* Pre-menopause
* Obese with a BMI between 30 kg/m2 and 40 kg/m2
* Has been obese for at least one year prior to screening
* Non-lactating
* Non-pregnant; has a negative urine pregnancy test result, does not plan on becoming pregnant during the study be willing to continue to practice appropriate birth control (such as implants, injectables, oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation, or a vasectomized partner) during the entire study duration.

Exclusion Criteria:

* Has obesity of known endocrine origin (e.g., Cushing's disease, Addison's disease, hypothalamic tumor);
* Has a medical history (e.g., morbid childhood obesity) and/or physical characteristics (e.g., polydactyly) suggestive of genetic obesity (e.g., ob/ob genotype) or syndromatic obesity (e.g., Prader-Willi syndrome, Bardet Biedl syndrome);
* Previous surgical procedures for weight loss;
* Has had liposuction within 1 year before screening or is planning to have liposuction during the study;
* History of bulimia or evidence of laxative abuse;
* Has had a body weight loss of more than 4 kg in the 90 days prior to screening;
* Has taken drugs capable of influencing body weight 30 days prior to screening;
* Has recently (<6 months prior screening) started or plans on starting a smoking cessation program;
* Has had a major change in daily physical activity (e.g., initiation of an exercise program) or started a weight loss program within 90 days prior to screening;
* Has a clinically significant history or presence of any of the following conditions:

  * Active or past history of cardiovascular or cerebrovascular disease including unstable angina, myocardial infarction, transient ischemic attacks/stroke, clinically significant arrhythmia, congestive heart failure, or cardiac valve abnormalities;
  * Type 1 diabetes mellitus;
  * Type 2 diabetes mellitus on treatment other than metformin monotherapy and/or diet with HbA1c >8%;
  * Severe type 2 diabetes with history of ketoacidosis or diabetic ulcers, or presence of retinopathy, neuropathy, or nephropathy;
  * Renal insufficiency defined as a serum creatinine equal or higher than 1.5 mg/dL (133 µmol/L) at screening;
  * Malignant disease within 5 years of screening;
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) higher than 2 x ULN;
  * Thyroid-stimulating hormone (TSH) outside of the normal range;
* Plans on having any surgery (elective or otherwise) during the course of the study;
* Has uncontrolled hypertension (sitting blood pressure >160/95 mmHg at screening or randomization), uncontrolled hyperlipidemia (triglycerides [TG] >400 mg/dL or low-density lipoprotein cholesterol [LDL-C] >190 mg/dL), or uncontrolled diabetes (HbA1c >8%);
* History of asthma;
* History of peptic ulcers associated with gastrointestinal bleeding or that required treatment with H2 blockers or proton pump inhibitors in the last 12 months.
* Has undergone bilateral Ovarectomy.
* History of HIV
* Has clinical laboratory test values (chemistry, hematology, or urinalysis) judged to be clinically significant by the investigator;
* Has a physical examination or electrocardiogram (ECG) with significant abnormalities, as judged by the investigator;
* Currently abuses drugs or alcohol or has a history of abuse that in the investigator's opinion could cause the subject to be noncompliant with study procedures;
* Has psychiatric or neurological disorders requiring chronic medications (e.g., antidepressants) and/or subjects score of > 8 on The Harvard Department of Psychiatry and National Depression Screening Day Scale (THE HANDS) (meaning " Presence of a major depressive episode is likely.").
* Chronic or as needed use of antihistamines;
* Has not been on a stable treatment regimen with any of the following medications for a minimum of 90 days prior to screening:

  * Oral contraceptives;
  * Antihypertensive agents;
  * Metformin;
  * Lipid-lowering agents; or
  * Thyroid replacement therapy;
* Has been treated over the past 60 days, is currently treated, or is expected to require or undergo treatment with any of the following excluded medications;

  * All prescription or over-the-counter agents taken for the purpose of weight reduction, including (but not limited to) the following anti obesity agents:

    * Prescription drugs such as orlistat, sibutramine, rimonabant and phentermine;
    * Over-the-counter antiobesity agents (e.g., herbal supplements or other alternative remedies);
  * Psychotropic/neurological agents including the following:

    * Antipsychotic agents (e.g., olanzapine, clozapine, risperidol, lithium, etc.).
    * Antiepileptic agents (e.g., topiramate , zonisimide, valproate, carbamazepine);
    * Antidepressant agents including the following: monoamine oxidase inhibitors, bupropion, tricyclic antidepressants, and tetracyclic antidepressants; and selective serotonin reuptake inhibitors (e.g., Fluoxetine, bupropion);
  * Systemic steroids administered by oral, intravenous, or intramuscular route;
  * Drugs that directly affect gastrointestinal motility (e.g., metoclopramide, and chronic [taken for more than 10 days within a 6- month period] macrolide antibiotics such as erythromycin and newer derivatives);
  * Calcitonin;
  * Insulin;
  * Exenatide;
  * Sulfonylureas;
  * Meglitinides
* Has received any investigational drug within 90 days of screening;
* Receipt of any investigational treatment (drug or device) within 90 days prior to screening;
* Is an immediate family member of personnel directly affiliated with the study at the investigative site, or is personally directly affiliated with the study at the investigative site; or
* Is employed by OBEcure Ltd.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 187 (Actual)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
change in body weight in Kg or % of initial body weight and/or proportion of subjects achieving > 2.5% and/or >5.0 % weight loss. | From baseline to week 12

SECONDARY OUTCOMES:
Change in obesity associated conditions | from baseline to Week 12
Safety parameters | From baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Yaffa Beck, PhD, CEO, Study Director — OBEcure Ltd.; Luc Van Gaal, MD Professor, Principal Investigator — UZ Antwerpen; Nir Barak, MD, Study Chair — OBEcure Ltd.
Locations (12):
- Belgium (4):
  - GP: Dr. Van Mulders, Aalst
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Germany (2):
  - Zentrum für Therapiestudien, Leipzig
  - CRS Clinical Research Services, Mönchengladbach
- Netherlands (6):
  - Emotional Brain, Almere Stad
  - GP: Dr. Rol, Bennebroek
  - Wecor, Etten-Leur
  - PT&R, Geleen
  - AMWO, Rotterdam
  - AMWO, The Hague